CLINICAL TRIAL: NCT05125263
Title: Comparison of the Effects of Kinesio Taping and Mulligan Taping on Patellofemoral Pain Syndrome.
Brief Title: Effects of Kinesiotaping and Mulligan Tapping on PFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00943 Zainab Tariq
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; Range of motion; Kinesiotaping; Mulligan taping; Physical performance measure
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): This group receives KinesioTaping along with conventional treatment
  Interventions: Other: kinesiotaping group
- group 2 (Experimental): This group receives mulligan taping along with conventional treatment
  Interventions: Other: mulligan taping group

INTERVENTIONS:
Other: kinesiotaping group — Kinesio-taping with conventional therapy 24, 48 and 72 hours standardized therapeutic KT application along with conventional therapy (hot pack, strengthening and stretching exercises). The patient laid supine.To maintain proprioceptive stimulation in the quadriceps (from origin towards insertion) and to alleviate the tension of hamstring muscle, a 'Y'-shaped kinesiotaping will be applied. Afterward, 2 pieces of 'I'-shaped tapes were stretched by 75% through the mechanical correction technique and will be applied around the patellar circumference in the way that it would allow the patella to move naturally in the femoral cavity while the knee was in 45 flexion
  CONVENTIONAL THERAPY:
  Stretching of hamstrings 10 reps 10 sec hold. Straight leg raise 3 sets* 10 reps, 1 min interval. Strengthening of Quadriceps (quads isometric) and VMO with 10 reps and 3 sets, 1 min interval) Squatting (10 reps* 3 sets, 1 min interval)
  Arms: group 1
Other: mulligan taping group — Mulligan taping will be applied while patient in standing position and the hip, knee will be internally rotated and flexed to 20 degree. Rigid tape will be applied from neck of fibula which will be passing anteriorly over the tibia to secure internal rotation of tibia at the knee, and passing below the medial joint line and behind the knee, 2 superimposed layers of 38-mm rigid tape will be applied in a spiral fashion. Tape will be applied for 24, 48 and 72 hours. And it must come off immediately if any pain and skin irritation is experienced. Along with conventional therapy.
  Stretching of hamstrings 10 reps 10 sec hold. Straight leg raise 3 sets* 10 reps, 1 min interval. Strengthening of Quadriceps (quads isometric) and VMO with 10 reps and 3 sets, 1 min interval) Squatting (10 reps* 3 sets, 1 min interval)
  Arms: group 2

SUMMARY:
The aim of this research is to compare the effects of kinesiotaping and mulligan taping on pain, hamstring flexibility, cadence and physical performance of lower limb in patients suffering from patellofemoral pain syndrome according to time duration 24, 48 and 72 hours. Randomized controlled trial done at Riphah International University Rawalpindi campus, Pakistan Railway Hospital and private clinics of twin cities. The sample size was 20. The subjects were divided in two groups, 10 subjects in kinesiotaping group and 10 in mulligan taping group. Study duration was 1 year. Sampling technique applied was non probability convenient sampling technique. Both males and females of 20-35 age bracket having anterior knee pain for more than 2 months and ≥3 pain on NPRS while performing activities i.e. ascending descending stairs, squatting and sitting for extending periods of time were included in study. Tools used in study are NPRS, Kujala pain rating sale, goniometer, active knee extension test, time up and go test.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a frequent musculoskeletal pathology affecting population like adults, teenage boys/girls, military and athletic individuals. It is a probable reason for anterior knee pain in individuals, also known as runner's knee. It is mainly defined as the individuals experience anterior knee pain, including other structural pathology like of patella and retinaculum. There is no related problem of intra articular and peri-patellar impairments. The causes of PFPS includes muscular imbalance of vastus lateralis and vastus medialis, maltracking of patella, instability of hip joint and hind most foot eversion. According to literature the PFPS is mostly common in active young population along with that women are more prone to develop this disease condition as compare to males because of their pelvis anatomy. Wider pelvis area in women causes more stress on knees. The reason of knee joint pain in older people is arthritis (age related degenerative changes). KT tapping has elastic properties like skin, stretching 30 % to 40 % stretching lengthwise. KT has water proof qualities and can be applied for 3 to 5 days. By applying KT over the skin of affected muscle or on joint surface, it reduces the pain, improves the circulation by giving positional impulse through skin, and modify interstitial tissue to reduce skin tension. Mulligan introduced a tapping technique called Mulligan tapping along with Mobilization with Movement technique development. Mulligan tape method prevents the positional malalignment in the joint. Tape may be applied for a week or two and not cause any harm along with mobilization Literature review: Anne Hickey et al. conducted a study in Australia in 2016. In this study effects of mulligan knee tapping technique on pain and lower limb biomechanics was determined. The study concluded that the technique successfully reduced the knee pain, decreased hip internal rotation and active gluteal muscles earlier. Leticia Lopes Aguiar et al. conducted a study in which he determines the effect of mulligan concept among ballet dancers. The study concluded that mulligan concept had significant results to improve pain threshold. Samara Alencar Melo et al. in which KT taping effects was determined on pain and muscular performance in patellofemoral pain syndrome patients did a study in 2018. In this RCT, the results showed that KT causes reduction in pain within 72 hours after its application without causing tension around skin. In 2017, Neelam Rehman et al. in Pakistan conducted a study. In this research the immediate effects of KT on pain in athletic population having PFPS was determined. The study concluded that KT had immediate effects in reducing pain and it can be used to treat immediate post injuries in athletic population.

ELIGIBILITY:
Inclusion Criteria:

* Anterior knee pain which is persisting longer than two months (pain on ascending and/or descending stairs, squatting, sitting for extended periods of time).
* Pain scoring rate on NPRS scale three or more during at least two activities.
* Age between 20 and 35 years.
* Both Male and female.

Exclusion Criteria:

* Meniscus tears, bursitis, patellar tendon, any ligamentous injury, any joint degeneration changes and patellofemoral dislocation and/or frequent subluxation.
* Undergone lower extremity surgery
* Patients having knee pain due to hip, lumbar spine and ankle joints
* Dermatitis and any other skin problem

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Kujala pain Rating score | 72 hours
  The Kujala pain rating scale is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. For example, a 'Limp' score would be scored as follows: none (5), slight/periodic (3), constant (0). Total scores range from 0 to 100.

SECONDARY OUTCOMES:
Numeric pain rating scale | 72 hours
  Numeric pain rating scale is used to assess the intensity of pain before and after intervention. Its value ranges from 0-10. O indicates no pain and 10 indicate maximum pain. Reliability of this tool is r=0.957. It will be measured at 24 hour, 48 hour, and 72 hour.
Time Up and Go | 72 hours
  Time up and go test is used to assess the dynamic balance ability, in this subject took to rise from 46cm height arm chair, walk 3 meter, turn back at affected side and walk back to chair and sit. Reliability of this tool is r = 0.98 to 0.99. It will be measured at 24 hour, 48 hour, and 72 hour
Active Knee Extension Test | 72 hours
  To check hamstring flexibility, patient position is in supine and effected leg is in 90-degree hip flexion. Patient is asked to extend the knee. The actual cutoff value for the Active knee extension test is 160. Normal individual has range of >160 or equal to160 (=160) and angle <160 considered hamstring tightness.)

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No